CLINICAL TRIAL: NCT01424358
Title: Web-based Education on Oral Cancer for Primary Care Physicians in Ohio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Model: Parallel | Masking: Single
Other Study IDs: 11-16008; 7K23DE016890-07 (NIH)
Record Dates: First submitted 2011-08-22; First posted 2011-08-29 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2012-12

CONDITIONS: Oral Cancer
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Web-based Educational (Experimental)
  Interventions: Other: Web-based Educational Intervention

INTERVENTIONS:
Other: Web-based Educational Intervention — The intervention group will be invited to participate in the web-based educational program. PCPs in the intervention group will be asked to view the educational module which will be followed by an assessment. This group will be tested on the following knowledge outcomes: Index of knowledge of risk factor for oral cancer and Index of knowledge of diagnostic procedures for oral cancer.

SUMMARY:
Objective:

The experimental design is a one-site, randomized experimental web-based educational feasibility intervention trial, with approximately 50% primary care physicians (PCPs) in the intervention group and approximately 50% PCPs on the control group, giving a total of 159 participants. All 159 participants have willingly provided their e-mail addresses, as part of a survey they previously completed entitled, "Survey of Health Professionals on Oral Cancer in Ohio- Intervention to Prevent Delayed Diagnosis of Oral Cancer."

DETAILED DESCRIPTION:
The main specific aim is to determine the short-term effectiveness of a web-based educational intervention for primary care physicians (PCPs) in Ohio to improve the following:Index of knowledge of risk factors for oral cancer, and Index of knowledge of diagnostic procedures for oral cancer

The following hypothesis will be explored: The use of a web-based educational module for PCPs in Ohio regarding oral cancer will increase the proportion of the PCPs in the high score category for the following indices: Index of knowledge of risk factors of oral cancer, and Index of knowledge of diagnostic procedures for oral cancer

ELIGIBILITY:
Inclusion Criteria:

* The PCP's who participated in Specific Aim #2 (Survey of Healthcare Professionals on Oral Cancer in Ohio ) of the NIH K23 grant proposal, "Intervention to Prevent Delayed Diagnosis of Oral Cancer", will be eligible to participate in this Web-Based Education on Oral Cancer.
* Possessing the ability to give voluntary consent to participate. Participating in the web-based educational intervention is am implication of consent.
* All participants are expected to be relatively healthy.

Exclusion Criteria:

• Unable to have access to the internet to be able to participate in the web-based education.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Index of knowledge of diagnostic procedure for oral cancer | An average of 8 months from the time of the initial email sent on 7/21/11.
  The list of participants will be sent an initial email inviting them to view the module and complete a pre test (control group) or a post test (intervention group). Reminder emails will be sent every 2 months for up to 6 months following the initial email. It is expected that at least a 15% higher proportion of Intervention group PCPs will attain the high score category for each of this index, as compared to the Control group PCPs.

SECONDARY OUTCOMES:
To determine if a change in Stage of Diagnosis of Oral Cancer occurred for the particular year of Web-based Educational Intervention. | 3 years
  Three years post-web-based education intervention data will be requested from Ohio Cancer Incidence Surveillance System (OCISS). OCISS's cleaning and processing of the data takes approximately three years. Comparison using Chi-square will be carried out pre- and post- intervention years.
Index of knowledge of risk factors for oral cancer. | An average of 8 months from the time of the initial email sent on 7/21/11.
  The list of participants will be sent an initial email inviting them to view the module and complete a pre test (control group) or a post test (intervention group). Reminder emails will be sent every 2 months for up to 6 months following the initial email. It is expected that at least a 15% higher proportion of Intervention group PCP's will attain the high score category for this index, as compared to the Control group PCP's.

CONTACTS AND LOCATIONS:
Overall Officials: Alvin G Wee, DDS, MS, MPH, Principal Investigator — Creighton University
Locations (1):
- Creighton University School of Dentistry, Omaha, Nebraska, United States

REFERENCES:
- [Background] Jemal A, Thomas A, Murray T, Thun M. Cancer statistics, 2002. CA Cancer J Clin. 2002 Jan-Feb;52(1):23-47. doi: 10.3322/canjclin.52.1.23. PMID 11814064
- [Background] Canto MT, Devesa SS. Oral cavity and pharynx cancer incidence rates in the United States, 1975-1998. Oral Oncol. 2002 Sep;38(6):610-7. doi: 10.1016/s1368-8375(01)00109-9. PMID 12167440
- [Background] Silverman S Jr. Demographics and occurrence of oral and pharyngeal cancers. The outcomes, the trends, the challenge. J Am Dent Assoc. 2001 Nov;132 Suppl:7S-11S. doi: 10.14219/jada.archive.2001.0382. PMID 11803655
- [Background] Mashberg A, Garfinkel L. Early diagnosis of oral cancer: the erythroplastic lesion in high risk sites. CA Cancer J Clin. 1978 Sep-Oct;28(5):297-303. doi: 10.3322/canjclin.28.5.297. No abstract available. PMID 100189
- [Background] Horowitz AM, Nourjah PA. Factors associated with having oral cancer examinations among US adults 40 years of age or older. J Public Health Dent. 1996 Fall;56(6):331-5. doi: 10.1111/j.1752-7325.1996.tb02460.x. PMID 9089528
- [Background] Canto MT, Drury TF, Horowitz AM. Use of skin and oral cancer examinations in the United States, 1998. Prev Med. 2003 Sep;37(3):278-82. doi: 10.1016/s0091-7435(03)00124-5. PMID 12914834
- [Background] Horowitz AM, Moon HS, Goodman HS, Yellowitz JA. Maryland adults' knowledge of oral cancer and having oral cancer examinations. J Public Health Dent. 1998 Fall;58(4):281-7. doi: 10.1111/j.1752-7325.1998.tb03010.x. PMID 10390710
- [Background] Goodman HS, Yellowitz JA, Horowitz AM. Oral cancer prevention. The role of family practitioners. Arch Fam Med. 1995 Jul;4(7):628-36. doi: 10.1001/archfami.4.7.628. No abstract available. PMID 7606301